CLINICAL TRIAL: NCT00976157
Title: Serial Changes of Soluble TREM-1 Level in Bronchoalveolar Lavage Fluid During Ventilator-associated Pneumonia
Brief Title: Serial Changes in sTREM-1 During Ventilator-associated Pneumonia (VAP)
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Cheng-Ho Tsai,superintendent, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-201
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Pneumonia
Keywords: STREM-1; BAL; VAP
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ventilator-associated pneumonia
  Interventions: Procedure: Bronchoscopy BAL

INTERVENTIONS:
Procedure: Bronchoscopy BAL — The bronchoscope was passed through endotracheal tube via a specific adaptor without topical anesthesia. The bronchoscope was introduced and wedged into the segmental bronchial orifice where pneumonia was suspected. Five aliquots of 20ml sterile saline were instilled and aspirated gently. The first aliquot was discarded and the last 4 aliquots were pooled for analysis. Part of the retrieved specimen in the first BAL fluid was sent to the laboratory immediately after collection for measurement of sTREM-1 level, the rest of sample was sent to microbiology lab for quantitative culture.

SUMMARY:
Triggering receptor expressed on myeloid cells (TREM)-1 is a recently described molecule that plays an important role in myeloid cell-activated inflammatory responses. The aim of this study was to investigate the evolutional change of soluble TREM-1 (sTREM-1) in bronchoalveolar lavage (BAL) fluid of clinically diagnosed ventilator-associated pneumonia (VAP) and its correlation with response to treatment and outcome.

DETAILED DESCRIPTION:
A prospective, interventional study conducted between August 2006 and August 2007 in MICU in Mackay Memorial Hospital, 35 patients with clinically diagnosed VAP were investigated. sTREM-1 was measured in BAL samples using ELISA at the onset, 4th - 5th and 7th - 9th day of clinical diagnosis of VAP.Of these 35 patients, 27 had positive BAL culture. The sTREM-1 levels in BAL fluid were measured and compared between patients with positive BAL culture and negative BAL culture. Serial changes in sTREM-1 levels were evaluated in relation to patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (older than 18 years)with clinically suspected VAP

Exclusion Criteria:

* mechanically ventilated patients post cardiopulmonary resuscitation
* patients with end stage diseases with life expectancy less than 3 months
* patients with solid or hematology transplantation
* patients on immunosuppressive agents

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were clinically suspected to have VAP were enrolled in the study. VAP was clinically diagnosed with a new infiltrate on a chest radiograph in a patient receiving mechanical ventilation for more than 48 hr with at least one of the following: purulent tracheal secretions, a body temperature >38°C or <36°C, and leukocytosis (WBC > 10,000/mm³) or leukopenia (WBC < 4000/mm³)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
mortality | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Chien Liang Wu, MD, Principal Investigator — Mackay Memorial Hospital, Taipei, Taiwan
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan